CLINICAL TRIAL: NCT01305590
Title: Understanding Medication Adherence Among HIV Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Bureau of Economic Research, Inc. (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 0004; P01AG005842 (NIH)
Record Dates: First submitted 2010-11-30; First posted 2011-02-28 (Estimated); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Patient Commitment Preferences for Medication Adherence
Keywords: HIV; AIDS; Medication Adherence; Commitment Devices; Behavioral Economics
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Medication Adherence

STUDY DESIGN:
Intervention Model Description: We will survey participants to see if they would prefer more commitment, in the form of a "Take-Medication-Get-Paid" plan; less commitment, in the form of an "Attend-Clinic-Get-Paid" plan; or if they would prefer to designate their own levels of commitment.
  The study also included 70 individuals in a passive control (PC) arm, who did not receive financial incentives. Individuals in the PC arm were not enrolled in the randomized trial but met basic study eligibility criteria during the same time period.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Survey (Other): We will survey participants to see if they would prefer more commitment, in the form of a "Take-Medication-Get-Paid" plan; less commitment, in the form of an "Attend-Clinic-Get-Paid" plan; or if they would prefer to designate their own levels of commitment.
  Interventions: Other: Survey to Understand Medication Adherence among HIV Patients

INTERVENTIONS:
Other: Survey to Understand Medication Adherence among HIV Patients — We want to better understand how this particular population would react to commitment devices designed to increase medication adherence. We will survey participants to see if they would prefer more commitment, in the form of a "Take-Medication-Get-Paid" plan; less commitment, in the form of an "Attend-Clinic-Get-Paid" plan; or if they would prefer to designate their own levels of commitment.

SUMMARY:
In anticipation of a pilot study incorporating behavioral economics into the treatment of infectious diseases, we will conduct a survey with HIV/AIDS patients at the Ponce Clinic (Infectious Disease Program of Grady Memorial Hospital, Emory University School of Medicine, Atlanta, GA).

DETAILED DESCRIPTION:
We are planning a study to improve health outcomes among patients with HIV/AIDS using insights from behavioral economics and financial incentives. We will conduct a survey with HIV/AIDS patients at Ponce Clinic (Infectious Disease Program of Grady Memorial Hospital, Emory University School of Medicine, Atlanta, GA). The patients will be low-income persons living with HIV/AIDS and possessing varying degrees of medication adherence. We want to better understand how this particular population would react to commitment devices designed to increase medication adherence. We will survey participants to see if they would prefer more commitment, in the form of a "Take-Medication-Get-Paid" plan; less commitment, in the form of an "Attend-Clinic-Get-Paid" plan; or if they would prefer to designate their own levels of commitment.

ELIGIBILITY:
Inclusion Criteria:

* HIV/AIDS patients currently receiving treatment at the Ponce Clinic at the Infectious Disease Program of Grady Memorial Hospital (Emory University School of Medicine).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2011-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Commitment Preferences for Increasing Medication Adherence | Up to 4 months
  We will measure whether participants prefer more commitment, in the form of a "Take-Medication-Get-Paid" plan; less commitment, in the form of an "Attend-Clinic-Get-Paid" plan; or if they would prefer to designate their own levels of commitment.

SECONDARY OUTCOMES:
Medication Adherence and Commitment Preference | Up to 4 months
  We will measure how subjects' medication adherence affects their stated commitment preferences.

CONTACTS AND LOCATIONS:
Overall Officials: David I Laibson, Ph.D, Principal Investigator — National Bureau of Economic Research
Locations (1):
- Ponce Clinic, Emory University School of Medicine, Atlanta, Georgia, United States

REFERENCES:
- [Result] Alsan M, Beshears J, Armstrong WS, Choi JJ, Madrian BC, Nguyen MLT, Del Rio C, Laibson D, Marconi VC. A commitment contract to achieve virologic suppression in poorly adherent patients with HIV/AIDS. AIDS. 2017 Jul 31;31(12):1765-1769. doi: 10.1097/QAD.0000000000001543. PMID 28514277